CLINICAL TRIAL: NCT02119949
Title: A Randomized Double-blind Placebo-controlled Trial to Working Memory Training in Substance Abusers
Brief Title: Working Memory Training for Substance Dependent Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Ingmar Franken, Professor, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2014-04-08; First posted 2014-04-22 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Substance Dependency; Addiction; Anxiety; Depression
Keywords: Substance abuse; Addiction; Working memory; Craving; Impulsivity; Attention control
MeSH Terms: conditions — Behavior, Addictive; Anxiety Disorders; Depression; Substance-Related Disorders; Impulsive Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Working memory training (Experimental)
  Interventions: Behavioral: Working memory training
- Placebo training (Placebo Comparator)
  Interventions: Behavioral: Placebo training

INTERVENTIONS:
Behavioral: Working memory training — The working memory training started the day after the pre-test and included 24 sessions of 25 minutes each. Participants trained, under supervision of an experimenter, on weekdays in the clinic. The training consisted of two tasks: the Symmetry Span and the N-back Task. Participants in the experimental group executed versions of these task that adapt to their working memory capacity, to train their working memory optimally.
  Arms: Working memory training
Behavioral: Placebo training — The working memory training started the day after the pre-test and included 24 sessions of 25 minutes each. Participants trained, under supervision of an experimenter, on weekdays in the clinic. The training consisted of two tasks: the Symmetry Span and the N-back Task. Participants in the placebo group executed easy versions of these task that did not adapt to their level, to prevent training.
  Arms: Placebo training

SUMMARY:
Background: Substance abusers show impaired working memory (WM) functioning. Promising findings show training WM results in an improved working memory capacity (WMC) and a decrease of clinical symptoms in a range of disorders, including alcohol addiction.

Aim: To test the effect of a WM training in addition to treatment as usual (TAU) on substance use, craving, WMC, impulsivity, attention bias and psychopathology.

Design: A randomized double-blind placebo-controlled trial with a parallel group design. The WM training adapted to participants' WMC whereas the placebo training consisted of non-adaptive easy versions of these tasks.

Setting: Two departments of an addiction treatment clinic in Rotterdam, the Netherlands.

Participants: 120 inpatients diagnosed with an alcohol, cannabis or cocaine dependency who were in treatment as usual .

Measurements: Primary outcome measures: Substance use and craving. Secondary outcome measures: WMC, impulsivity, attention bias and psychopathology. Participants were assessed before and after 24 sessions of WM training as well as two months after the training.

ELIGIBILITY:
Inclusion Criteria:

* Substance dependency: cocaine, cannabis or alcohol

Exclusion Criteria:

* Age below 16 or above 67
* Current psychosis
* Neurological complaints

Ages: 16 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Craving: Desires for Alcohol Questionnaire and Desires for Drug Questionnaire score change and Obsessive Compulsive Drug Use Scale and Obsessive Compulsive Drinking Scale score change between pre and post training and follow up (two months after post) | Pre (baseline), post (after 4 weeks of training-starting 1 day after pre-test) and follow-up (2 months after post-test)
  The 14-item Desires for Drug Questionnaire (DDQ) and the 13-item Desires for Alcohol Questionnaire (DAQ) measure instant craving to respectively drug and alcohol. The DDQ is based on the DAQ.
  The Obsessive Compulsive Drug Use Scale (OCDUS) and Obsessive Compulsive Drinking Scale (OCDS) measure the subjective interference and distress caused by respectively drug and alcohol related thoughts and compulsive-behavior patterns.

SECONDARY OUTCOMES:
Change in Digit Span score on pre and post training and follow up after two months | Pre (baseline), post (after 4 weeks of training-starting 1 day after pre-test) and follow-up (2 months after post-test)
  The Digit Span task consists of two parts: the forward Digit Span is a frequently used measure for short term memory, an important subcomponent of the memory system (Shipstead, Redick, & Engle, 2012) and the backward version measures WM.
Change in Reading Span partial-scredit uni score on pre and post training and follow up after two months | Pre (baseline), post (after 4 weeks of training-starting 1 day after pre-test) and follow-up (2 months after post-test)
  The Reading Span measures the processing and storage functions of WM (Shipstead et al., 2012), specifically participants' ability to shift between two tasks and to cope with proactive interference.

OTHER OUTCOMES:
Change in Barratt Impulsivity Scale-11 score on pre and post training and follow up after two months | Pre (baseline), post (after 4 weeks of training-starting 1 day after pre-test) and follow-up (2 months after post-test)
  The 30-item Barratt Impulsivity Scale-11 (BIS-11) measures impulsivity.
Change in Stroop score on pre and post training and follow up after two months | Pre (baseline), post (after 4 weeks of training-starting 1 day after pre-test) and follow-up (2 months after post-test)
  The Stroop measures participants' attention bias for addiction related stimuli.
Change in Beck Depression Inventory - Second Edition (BDI-II) score on pre and post training and follow up after two months | Pre (baseline), post (after 4 weeks of training-starting 1 day after pre-test) and follow-up (2 months after post-test)
  The Beck Depression Inventory - Second Edition (BDI-II) measures the severity of depression in 21 statements, with four levels of increasing severity each.
Change in State-Trait Anxiety Inventory (STAI) score on pre and post training and follow up after two months | Pre (baseline), post (after 4 weeks of training-starting 1 day after pre-test) and follow-up (2 months after post-test)
  The State-Trait Anxiety Inventory (STAI) measures self-reported anxiety in 40 questions on a 4-point scale. The questionnaire consists of two parts; state and trait anxiety, respectively transient and dispositional anxiety.
Change in substance use, measured with the Addiction Severity Index over pre-, post (1 day after training) and follow-up (2 months after post-test) measurements. | Pre (baseline), post (after 4 weeks of training-starting 1 day after pre-test) and follow-up (2 months after post-test)
  The Addiction Severity Index (ASI) is a semi-structured interview that measures the severity of addiction in 25 questions concerning seven problem areas: medical problems, employment problems, drug use, alcohol use, family and social problems, criminality, and psychiatric problems. We used three of these questions to assess the severity of participants' abuse problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Bouman Clinic, Rotterdam, South Holland, Netherlands